CLINICAL TRIAL: NCT06172491
Title: Harnessing the Power of Technology to Transform Delirium Severity Measurement in the ICU
Brief Title: Automating Delirium Severity in the ICU
Acronym: ADS-ICU
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Heidi L. Lindroth PhD RN, Heidi L. Lindroth, Ph.D., Nurse Scientist, Assistant Professor of Nursing, Mayo Clinic
Other Study IDs: 22-003098
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Intensive Care Unit Delirium; Encephalopathy; Delirium
Keywords: Delirium; Severity; Digital marker; Computer Vision; Artificial Intelligence
MeSH Terms: conditions — Brain Diseases; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No Delirium Severity: Patients who did not experience a level of delirium severity (subsyndromal, mild, moderate, severe)
- Delirium Severity: Patients who did experience a level of delirium severity (subsyndromal, mild, moderate, severe)

SUMMARY:
The goal of this observational study is to develop a passive digital marker (PDM) for delirium severity and examine its performance in comparison to validated delirium severity tools in ICU patients >50 years of age.

The main questions it aims to answer are:

* Is the trained convolutional neural network able to reliably measure delirium severity.
* Is the Passive Digital Marker able to accurately measure delirium severity
* Is the Passive Digital Marker acceptable and usable by frontline ICU nurse clinicians, patients, and their identified proxies (i.e., caregivers).

Participants will:

* Study participation involves a video camera recording you 24 hours per day while you are a patient in the Intensive Care Unit (ICU).
* Study staff will visit you 4 times each day you are in the ICU. You will be asked questions each time they visit to train the digital marker and see differences between assessments and camera data.

DETAILED DESCRIPTION:
Bedside cameras will stay up for at least 72 hours (about 3 days), it may be longer if delirium is being experienced and if the patient and or LAR (Legally Authorized Representative) agree to the cameras' continued recording.

The study team will come and ask the patient questions 4 times daily. We will ask questions about their general, mental, and emotional health, their mood and memory. During these visits, the study team will check the alertness of the patient. Alertness will be checked by voice; if they do not respond, we will tap their shoulder gently. We will ask the patient to do activities like remembering words and saying them back, shaking hands, and drawing an object or clock. The study team will administer assessments 4 times daily. Participants will be asked questions about their general, mental, and emotional health, as well as mood and memory. While performing these sessions, the study team will observe the level of awareness. Awareness will be assessed by voice; if they do not respond, we will have to do a gentle tap on their shoulders. The patient will be asked to perform activities such as: remembering words and repeating them back, handshaking, and drawing an object or clock.

In some cases, if the patient's level of awareness alertness is lowered, we will do observation only perform observation assessments. These assessments do not interfere with clinical care. Participation in this study is voluntary.

The study team will continue to follow the patient until discharged from ICU.

The bedside nurse, patient, or family can cover the cameras with a washcloth if needed for privacy. The faces of family and clinicians and the bathing suit areas of patients are blurred before analysis to protect privacy.

ELIGIBILITY:
Inclusion Criteria: • Age >50;

* Estimated length of stay >24 hours in ICU; and
* Are not admitted for acute alcohol intoxication, drug (prescribed or illicit) overdose or withdrawal.

Exclusion Criteria:

* Admitted for acute alcohol intoxication, drug (prescribed or illicit) overdose or withdrawal.
* Admitted for acute neuronal injury
* Unable to communicate with research team due to sensory deficits (aphasic, blind, deaf) or language (does not speak English)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Aging adults admitted to an intensive care unit
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2026-07-18 (Estimated); Study Completion 2026-12-18 (Estimated)

PRIMARY OUTCOMES:
Delirium Severity | 12-48 months
  The level of delirium severity will be measured by two types of prospective data collection. The first method is completed by study team members. A trained member of the study team will administer validated assessment tools 4xdaily from enrollment until ICU discharge or death. The Confusion Assessment Method for the Intensive Care Unit Severy Scale (CAM-ICU-7) is the gold standard for delirium severity measurement in the ICU. It is a 7-point scale, with 7 being severe delirium and 0 being no delirium. The second method is a passive digital marker (in development).
Acceptability of passive digital marker for delirium severity | 48 months - 60 months
  Participants and their identified care partners will be randomized 1:1 to either the Passive Digital Marker for Delirium Severity or usual care. The acceptability of the PDM by clinicians, patients, and care partners will be evaluated. The 4-question tool named Treatment Acceptability and Preference Questionnaire (TAPQ) is scored on a 5-point Likert scale. A higher score indicates higher acceptability.
Usability of passive digital marker for delirium severity | 48 months - 60 months
  Participants and their identified care partners will be randomized 1:1 to either the Passive Digital Marker for Delirium Severity or usual care. The usability of the PDM by clinicians, patients, and care partners will be evaluated. The 10-question System Usability Scale is scored on a Likert scale from 1-5. A higher score (0-100 range) indicates higher usability.

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raghu R, Nalaie K, Ayala I, Morales Behaine JJ, Garcia-Mendez JP, Friesen H, Leistikow K, Bhattacharyya A, Jayaraman A, Franco PM, Rabinstein A, Chlan LL, Boustani M, Herasevich V, Lindroth H. Harnessing the Power of Technology to Transform Delirium Severity Measurement in the Intensive Care Unit: Protocol for a Prospective Cohort Study. JMIR Res Protoc. 2025 Sep 25;14:e62912. doi: 10.2196/62912. PMID 40998312